Yelena Wu 

RAYS: Rural Youth and Adult Sun Protection Study

Version date: 12/3/24

# RAYS: Rural Youth and Adult Sun Protection Study (Community Members) Consent Cover Letter

## **SUMMARY**

- You are being asked to take part in a research study (RAYS). Your participation in this study is completely voluntary.
- The purpose of RAYS is to improve use of sun protective behaviors among youths living in rural communities in Utah and West Virginia.
- If you choose to participate in this study, you will be asked to complete a 30-minute interview about prevention efforts in your community regarding either injury prevention in sports or skin cancer prevention.
- This interview will take place by videoconference or telephone and will be recorded for quality control. The risks associated with study participation are minimal.
- If you decide you no longer want to participate in this study, you can contact us at any point and we will not collect any more information from you.
- We cannot guarantee any direct benefits to you, however, as compensation for your participation in the study you will receive \$20 for completing the study interview.

#### **BACKGROUND**

You are being asked to take part in a research study. Before you decide, it is important for you to understand why the research is being done and what it will involve. Please take time to read the following information carefully. Take time to decide whether or not to volunteer to take part in this research study.

The purpose of this study is to help prevent skin cancer. The goal of the study is to improve use of sun protective behaviors among youths living in rural communities in Utah and West Virginia. The lead investigators for this study are Dr. Yelena Wu from the University of Utah and Huntsman Cancer Institute, Dannell Boatman from West Virginia University and Dr. Kenneth Tercyak from the Lombardi Comprehensive Cancer Center at Georgetown University.

## **STUDY PROCEDURES**

We would like to learn what you know, think, and feel about protecting children in your community from skin cancer and ways to help them stay safe in the sun. We are also interested in your opinion about local efforts to educate members of your community about skin cancer and sun safety. If you choose to participate in this study, you will be asked to complete a 30-minute interview about these topics. This interview will take place by videoconference or telephone and will be recorded for quality control. You may be contacted about study activities via email, text messages, or phone calls.

## **RISKS**

The risk or discomforts associated with participating in this study are minimal. If you feel upset from any part of this experience, you can tell the researcher, who will tell you about resources available to help. Even though we do everything we can to protect the identity and privacy of participants, there is still a risk that data could be traced back to an individual. Once data is shared, participants can still request that their data be removed from data repositories. However, some data that have been distributed for approved research use cannot be retrieved.





Yelena Wu 

RAYS: Rural Youth and Adult Sun Protection Study

Version date: 12/3/24

## **BENEFITS**

While there are no direct benefits to you for participating in this study, you may gain awareness that you are contributing to new knowledge that may benefit others in rural communities who are at risk for skin cancer in the future.

## **PERSON TO CONTACT**

If there is anything that is not clear or if you would like more information, you can e-mail the research staff at <a href="mailto:rays.study@hci.utah.edu">rays.study@hci.utah.edu</a>. If you have any complaints or concerns about this study, you can contact Dr. Yelena Wu by leaving a message at (801) 585-9427. If you feel you have been harmed as result of participation, please call Dr. Yelena Wu at (801) 585-9427, who may be reached Monday through Friday, 8am-5pm.

**Institutional Review Board:** Contact the Institutional Review Board (IRB) if you have questions regarding your rights as a research participant. Also, contact the IRB if you have questions, complaints or concerns which you do not feel you can discuss with the investigator. The University of Utah IRB may be reached by phone at (801) 581-3655 or by e-mail at <a href="irb@hsc.utah.edu">irb@hsc.utah.edu</a>.

**Research Participant Advocate:** You may also contact the Research Participant Advocate (RPA) by phone at (801) 581-3803 or by email at <a href="mailto:participant.advocate@hsc.utah.edu">participant.advocate@hsc.utah.edu</a>.

## **VOLUNTARY PARTICIPATION**

If you change your mind, you can tell us anytime that you do not want to be in this study. We will not be able to collect new information about you, and you will be withdrawn from the research study. However, we can continue to use information we have already started to use in our research, as needed to maintain the integrity of the research.

# **COSTS AND COMPENSATION TO PARTICIPANTS**

There is no cost for participating in this study. You will be compensated up to \$20 for your participation in completing the study interview. Compensation will be provided to you directly following the study interview that you complete. Compensation will come in the form of cash-equivalent gift cards that may be physical or digital; if digital, this gift card will be issued to you by email.

# **CONFIDENTIALITY**

We will share information that identifies you with our research team members at the University of Utah at Huntsman Cancer Institute, Georgetown University at Lombardi Cancer Institute, West Virginia University, the National Cancer Institute (the study sponsor), and the University of Utah Institutional Review Board (IRB), which reviews research involving people to make sure the study protects your rights. Data will only be used for the present study and will not be saved and stored for future research. We will be video and/or audio recording the post-study interviews for feedback on participants' experience. All recordings and transcriptions will be stored in a secure manner. We will do everything we can to keep your information private but we cannot guarantee this. Study information will be kept in a secured manner and electronic records will be password protected. Your data will only be used for the present study and will not be saved or shared for future research.





Yelena Wu 

RAYS: Rural Youth and Adult Sun Protection Study

Version date: 12/3/24

## **CONSENT**

I confirm I have read the information in this consent form and have had the opportunity to ask questions. By participating in the interview, I agree to participate in this research. I will be provided with a copy of this form for my records.

I agree to take part in this research study as you have explained in this document.

We may contact you about future research that may be of interest to you or for other matters related to this study.

We greatly appreciate you participating in our study.

